CLINICAL TRIAL: NCT05930834
Title: Exercise Training and Adipose Tissue Insulin Sensitivity
Brief Title: Exercise Training and Insulin Sensitivity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: student collecting data not available
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, Professor and Interim Chair, Nutrition and Exercise Physiology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2096068
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): All subjects will undergo exercise training for 4 wks. 45-60 min of exercise, 4 sessions/wk supervised, 1 session unsupervised. intensity 60% of VO2 max
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — All subjects will undergo exercise training for 4 wks. 45-60 min of exercise, 4 sessions/wk supervised, 1 session unsupervised. intensity 60% of VO2 max

SUMMARY:
Regular exercise participation is known to reduce cardiometabolic disease risk but the impact that exercise training has on adipose tissue (AT) metabolism is poorly understood, particularly in humans. It is well established that exercise training improves whole-body glucose levels and increases insulin sensitivity, and this can occur within one or two weeks. These effects are usually due to adaptations in skeletal muscle, the tissue responsible for the majority of glucose disposal. However, many studies have now determined that exercise training also results in adaptations in AT that improve whole-body metabolic health by improving glucose uptake into the AT.

Skeletal muscle is thought to account for approximately 75-85% of glucose uptake , and this process is impaired in .individuals who are insulin-resistant state. It is postulated that the increased level of adiposity that accompanies severe obesity would result in higher dependency on AT for glucose uptake as the AT would be a bigger "sink". Thus the role of AT in inducing whole body insulin resistance is still unclear, particularly in individuals with obesity.

This study will examine the changes in AT glucose uptake before and after 4 weeks of exercise training in obese individuals and establish if there are sex differences.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers, weight stable (<4 kg) within the last 6 months will be recruited for this study.
* sedentary (not engaged in planned physical activities and performing less than a total of 2 h of physical activity per week during the last 6 months) men and women whose BMI is classified as obese (>30 kg/m2).

Exclusion Criteria:

* cardiovascular disease, uncontrolled hypertension (no beta blockers), smokers, pregnant, have any recent changes in hormonal birth control, or on any medications known to impact metabolism.
* All participants will be regular sleepers with a duration of 7-9 hours/night.
* Subjects with orthopedic limitations will not be included.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GLUT4 protein expression | 4 weeks
  protein expression
TB1CD4 protein expression | 4 weeks
  TB1CD4 protein expression

SECONDARY OUTCOMES:
percent body fat | 4 weeks
  Body fat will be measured using DEXA pre and post training

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Misouri, Columbia, Missouri, United States